CLINICAL TRIAL: NCT03111173
Title: Can Conventional ECG Technology Capture Fetal Cardiac Activity?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Martin Frasch, Research Assistant Professor, Obstetrics and Gynecology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00001556
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Fetal Monitoring
Keywords: ECG; Fetus; R peak extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Holter device (Other): Holter device to be attached to a Singleton or twin pregnant women at 32 weeks gestation to full term
  Interventions: Device: Holter Device

INTERVENTIONS:
Device: Holter Device — MyECG E3.80 Holter Recorder

SUMMARY:
This is a feasibility study for a new application for capturing fetal cardiac activity. The objective of this study is to determine if it is feasible to capture a fetal ECG signal using a Holter ECG device. As comparison we will use a standard Doppler Fetal Heart Rate (FHR) device.

DETAILED DESCRIPTION:
The objective of this study is to determine if it is feasible to capture a fetal ECG signal using a Holter ECG device. As comparison we will use a standard Doppler Fetal Heart Rate (FHR) device. To obtain the raw FHR data from this standard device we will use the currently approved "fetal EEG" monitor. The important distinction is that "fetal EEG" monitor will not be connected to fetal scalp electrode, but, rather, get the data from the regular, more routinely used and non-invasive Doppler FHR monitor. We expect that we will be able to validate our algorithm with our maternal and fetal ECG channels to derive the FHR.

We will attach a Holter ECG device (4 electrodes) and a standard Doppler FHR device to a pregnant woman who is between 32 weeks gestation and full term. ECG leads will be placed in four corners of the abdomen. The targeted length of the recording will be 30 minutes. The subject will remain supine and resting while the device is recording. Additionally, the recently approved fetal EEG monitor will be connected to the Doppler FHR device to allow us to obtain a "digital copy" of the standard FHR recording. We will do that in order to have the comparison during the offline processing of the abdominal ECG with regard to the location of the fetal R peaks. This procedure will be done after the subject's routine antepartum testing. No women in active labor will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Singleton or twin pregnant women at 32 weeks gestation to full term after routine antepartum testing.

Exclusion Criteria:

* None.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful extraction of fetal ECG from the maternal abdominal ECG signal | 12 months
  We will test the quality of correct identification of fetal R peaks of ECG from within maternal ECG signal by comparing the R-R-periods-derived instantaneous fetal heart rate (FHR) to the values determined by the standard-of-care ultrasound-derived FHR monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Martin G Frasch, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Efficient fetal-maternal ECG signal separation from two channel maternal abdominal ECG via diffusion-based channel selection Ruilin Li, Martin G. Frasch, Hau-tieng Wu (Submitted on 7 Feb 2017) There is a need for affordable, widely deployable maternal-fetal ECG monitors to improve maternal and fetal health during pregnancy and delivery. Based on the diffusion-based channel selection, here we present the mathematical formalism and clinical validation of an algorithm capable of accurate separation of maternal and fetal ECG from a two channel signal acquired over maternal abdomen. Subjects: Medical Physics (physics.med-ph); Data Analysis, Statistics and Probability (physics.data-an); Applications (stat.AP); Machine Learning (stat.ML) Cite as: arXiv:1702.02025 [physics.med-ph]
- See also: Efficient fetal-maternal ECG signal separation from two channel maternal abdominal ECG via diffusion-based channel selection — http://journal.frontiersin.org/article/10.3389/fphys.2017.00277/abstract